CLINICAL TRIAL: NCT07323355
Title: Effects of Single-Layer Versus Double-Layer Cesarean Scar Repair on Myometrial Thickness and Associated Clinical Outcomes
Brief Title: Single- vs Double-Layer Cesarean Scar Repair and Myometrial Thickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Didem Eşkin Tanrıverdi, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TABED 1-25-1872
Record Dates: First submitted 2025-12-03; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Caesarean Section; Cesarean Scar Closure; Cesarean Scar Defect (Isthmococele); Myometrial Thickness; Postpartum Complications; Clinical Outcomes
Keywords: Caesarean Section; Cesarean Scar Closure; Isthmococele; Myometrial Thickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-Layer Cesarean Scar Repair (Experimental): Participants in this arm receive double-layer closure of the cesarean section scar according to the study protocol. Outcomes such as myometrial thickness, scar integrity, and clinical parameters are measured. This arm is compared in parallel with the single-layer cesarean scar repair arm.
  Interventions: Procedure: Double-Layer Cesarean Scar Repair
- Single-Layer Cesarean Scar Repair (Experimental): Participants in this arm receive single-layer closure of the cesarean section scar according to the study protocol. Outcomes such as myometrial thickness, scar integrity, and clinical parameters are measured. This arm is compared in parallel with the double-layer cesarean scar repair arm.
  Interventions: Procedure: Single-Layer Cesarean Scar Repair

INTERVENTIONS:
Procedure: Double-Layer Cesarean Scar Repair — Participants in this arm undergo double-layer closure of the uterine incision during cesarean delivery. The procedure involves suturing the full thickness of the myometrium in the first layer, followed by a second continuous suture approximating the outer myometrium and serosa. Outcomes such as myometrial thickness, scar integrity, and clinical parameters are measured. This arm is compared in parallel with the single-layer cesarean scar repair arm.
  Arms: Double-Layer Cesarean Scar Repair
Procedure: Single-Layer Cesarean Scar Repair — Participants in this arm undergo single-layer closure of the uterine incision during cesarean delivery. The procedure involves a single continuous suture approximating the full thickness of the uterine wall. Outcomes such as myometrial thickness, scar integrity, and clinical parameters are measured. This arm is compared in parallel with the double-layer cesarean scar repair arm.
  Arms: Single-Layer Cesarean Scar Repair

SUMMARY:
Cesarean delivery (CD) is one of the most commonly performed surgical procedures worldwide, with a rising incidence particularly in high-income countries. Although often life-saving, cesarean delivery carries both short- and long-term maternal risks. Early complications include infection, hemorrhage, and thromboembolism, while inadequate uterine healing can lead to future complications such as uterine rupture and placenta accreta spectrum disorders. Additionally, cesarean scars may result in pregnancy complications, isthmocele formation, postmenstrual bleeding, pelvic pain, and dysmenorrhea. This highlights the need for optimization of the surgical technique. Despite increasing cesarean rates, there is no consensus on the optimal uterine closure method. Techniques vary in terms of the number of layers, suture locking style, and inclusion of the endometrium, and their comparative effectiveness in reducing scar defects remains unclear. Some previous studies have reported increased uterine rupture risk with single-layer locked sutures and better healing with double-layer closure, while others found no significant difference in scar outcomes. This study aims to investigate the effects of single- versus double-layer cesarean scar closure on myometrial thickness and its clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-44 years.
* Undergoing cesarean delivery at the study hospital's Obstetrics and Gynecology clinic.
* Evaluated as clinically eligible based on history, physical examination, abdominal ultrasonography, and routine preoperative laboratory tests, including:

Complete blood count (CBC), biochemical profile, prothrombin time (PT), activated partial thromboplastin time (aPTT), blood group determination. No abnormalities detected in the above assessments.

Exclusion Criteria:

- Presence of chronic diseases, including: Rheumatologic diseases, renal failure, vascular malformations, hypertension, cardiac disease, diabetes mellitus, obesity, thyroid disease, congenital hematologic disorders.

* Suspected or confirmed placenta previa or placenta accreta spectrum.
* Clinical chorioamnionitis.
* Anterior wall uterine myomas.
* History of low transverse nonstandard uterine incision.
* Predicted obstetric hemorrhage or other intraoperative complications.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study includes female participants only, as it investigates the effects of single-layer versus double-layer cesarean scar repair on uterine myometrial thickness and related clinical outcomes. Only women who are undergoing cesarean delivery and meet the inclusion criteria are eligible for participation.
Enrollment: 102 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Myometrial Thickness at Cesarean Scar Site | 6 months postoperatively
  Myometrial thickness at the cesarean scar site will be measured using transvaginal ultrasonography (TVUSG) by a qualified obstetrician at 6 months after surgery to compare the effects of single-layer versus double-layer cesarean scar closure.
  Measurement Tool / Parameter: TVUSG; residual myometrial thickness (mm). Units of Measure: Millimeters (mm).

SECONDARY OUTCOMES:
Cesarean Scar-Related Symptoms | 6 months postoperatively
  Presence of cesarean scar-related symptoms at 6 months after surgery. Parameters Assessed: Postmenstrual spotting (yes/no), pelvic pain (yes/no), dyspareunia (yes/no) Measurement Tool / Method: Clinical interview during follow-up visit and review of outpatient medical records.
  Units of Measure: Incidence (n, %)
Cesarean Scar Defect (Isthmocele) | 6 months postoperatively
  Presence of cesarean scar defect (isthmocele) detected by transvaginal ultrasonography.
  Measurement Tool / Method: Transvaginal ultrasonography. Units of Measure: Incidence (number of participants with isthmocele, %)
Major Uterine Scar-Related Complications | Up to 6 months postoperatively
  Occurrence of major uterine scar-related complications within 6 months after surgery.
  Parameters Assessed: Uterine rupture, cesarean scar pregnancy, abnormal uterine bleeding Measurement Tool / Method: Clinical examination and medical record review. Units of Measure: Incidence (n, %)
Morphological Characteristics of Cesarean Scar Defect | 6 months postoperatively
  Morphological characteristics of cesarean scar defect measured by transvaginal ultrasonography.
  Parameters Assessed: Isthmocele depth (mm), isthmocele width (mm) Measurement Tool / Method: Transvaginal ultrasonography. Units of Measure: Millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Merve Didem Eşkin Tanrıverdi, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Not Valid, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD are available which may be shared in necessary conditions.